CLINICAL TRIAL: NCT01627613
Title: Proof of Concept Study in Male and Female Intensive Care Patients to Investigate the Clinical Effect of Repetitive Orally Inhaled Doses of AP301 on Alveolar Liquid Clearance in Acute Lung Injury
Brief Title: Study in Intensive Care Patients to Investigate the Clinical Effect of Repetitive Orally Inhaled Doses of AP301 on Alveolar Liquid Clearance in Acute Lung Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apeptico Forschung und Entwicklung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP301-II-001; 2012-001863-64 (EudraCT Number)
Record Dates: First submitted 2012-06-20; First posted 2012-06-26 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Acute Lung Injury
Keywords: Peptide
MeSH Terms: conditions — Acute Lung Injury | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AP301 (Experimental): Treatment group
  Interventions: Drug: AP301
- saline solution (Placebo Comparator): Placebo group
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: AP301 — AP301 25 mg powder for reconstitution for solution for inhalation
  Orally delivered doses of 87.6 mg AP301 are inhaled every 12 hours (± 30 min), for a total of 7 days.
  Arms: AP301
Drug: Saline solution — Placebo solution (0.9% physiologic NaCl) is inhaled every 12 hours (± 30 min), for a total of 7 days.
  Arms: saline solution

SUMMARY:
The purpose of this study is to assess the effect of orally inhaled AP301 on alveolar liquid clearance in ALI (acute lung injury) patients with the purpose to assess the treatment associated changes of extravascular lung water (EVLW) within 7 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18
* intubated and mechanically ventilated male and female patients of the Intensive Care Units of the Department of Anesthesia, General Intensive Care and Pain Control
* meets the criteria of ALI (as defined by the American-European Consensus Conference on ALI/ ARDS):
* Onset of ALI within 48 hours
* Bilateral infiltrates seen on frontal chest radiograph
* PCWP ≤ 18 mm Hg or no clinical evidence of left atrial hypertension
* paO2/ FiO2 ratio ≤ 300 mm Hg
* EVLW in PiCCO® at screening ≥ 8 ml/PBW
* Meeting criteria for extensive hemodynamic monitoring according to investigators discretion
* ICU Patients being mechanically ventilated and are stable in this condition for at least 8 hours
* Negative pregnancy test and adequate contraception in female patients of childbearing potential
* Informed consent:
* For patients that are temporarily unable to consent (e.g. comatose patients) a subsequent informed consent has to be provided.

Exclusion Criteria:

* History of clinically relevant allergies or idiosyncrasies to AP301 or any other inactive ingredient(s) of the investigational product
* Brainstem death at screening
* Current evidence of septic shock as defined by the Surviving Sepsis Campaign (Presence of acute organ dysfunction secondary to infection plus hypotension with systolic blood pressure < 90 mm Hg or mean arterial pressure (MAP) < 70 mm Hg for not less than one hour which cannot be reversed with fluid resuscitation)
* Neutrophil count <0.3 x 109 L
* Patients under immunosuppression: high dose steroids (> 80 mg Prednisolone /d; > 300 mg hydrocortisone / d), cancer treatment (chemotherapy or biological) or therapy with other immunosuppressive agents for organ transplantation within 2 weeks
* BMI < 18.5 or > 35
* Cardiogenic pulmonary edema diagnosed by echocardiography or pulmonary artery catheter
* Pregnancy / lactation or intention to fall pregnant during the time course of the study
* Women of childbearing potential as well as men of procreative capacity who are not using adequate contraception
* Participation in other interventional drug trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
change in extravascular lung water within 7 days of treatment | change from baseline - day 7
  EVWL (measured with PiCCO® technique) until day 7 of treatment (AUC)

SECONDARY OUTCOMES:
Oxygenation index | baseline - day 7
  Oxygenation index (PaO2 / FiO2 ratio) until day 7 of treatment
ventilator plateau pressure | baseline - day 7
  Ventilator plateau pressure until day 7 of treatment
Murray Lung Injury Score | baseline - day 7
Ventilation parameters / lung function | baseline - day 7
Presence/absence/severity and duration of adverse effects - number and severity of adverse events (AEs), serious adverse events (SAEs) and suspected unexpected serious adverse events (SUSARs)) | baseline - day 7

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ullrich, Prof., Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Anesthesia, General Intensive Care and Pain Control,Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Krenn K, Lucas R, Croize A, Boehme S, Klein KU, Hermann R, Markstaller K, Ullrich R. Inhaled AP301 for treatment of pulmonary edema in mechanically ventilated patients with acute respiratory distress syndrome: a phase IIa randomized placebo-controlled trial. Crit Care. 2017 Jul 27;21(1):194. doi: 10.1186/s13054-017-1795-x. PMID 28750677